CLINICAL TRIAL: NCT02649543
Title: Comparison of Surgical Site Infection Rate Between Primary, Delayed Primary and Vacuum Assisted Closures. A Prospective Randomized Study.
Brief Title: Comparison of Surgical Site Infection Rate Between Primary, Delayed Primary and Vacuum Assisted Closures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eduardo Flores Villalba (Other)
Responsible Party: Sponsor-Investigator, Eduardo Flores Villalba, Associated investigator, Tecnologico de Monterrey
Organization: Tecnologico de Monterrey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACAB-01
Record Dates: First submitted 2015-11-25; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Surgical Wound Infection
Keywords: Surgical Wound Infection; Negative-Pressure Wound Therapy; Wound Closure Techniques; Laparotomy.; Abdominal Wound Closure Techniques
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Primary Closure (Active Comparator): Primary Closure is made after surgery.
  Interventions: Procedure: Primary Closure
- Delayed Primary Closure (Active Comparator): Delayed Primary Closure is made after at least 7 days.
  Interventions: Procedure: Delayed Primary Closure
- Vacuum Assisted Closure (Active Comparator): Vacuum Assisted Device is used in the wound.
  Interventions: Procedure: Vacuum Assisted Closure

INTERVENTIONS:
Procedure: Primary Closure — A double antibiotic scheme with a cephalosporin and metronidazole is used as prophylaxis, and the fascia was closed with a continuous Polyglycolic Acid 0 suture. Subcutaneous tissue was approximated with Polyglycolic Acid 3-0, and the skin is sutured using Polypropylene 2-0.
  Arms: Primary Closure
Procedure: Vacuum Assisted Closure — A double antibiotic scheme with a cephalosporin and metronidazole is used as prophylaxis, and the fascia is closed with a continuous Polyglycolic Acid 0 suture. The VAC® system is then used, with change of dressings every 48 hrs. The wound is closed using Polypropylene 2-0 only after healthy granulation tissue and no signs of infection are present.
  Arms: Vacuum Assisted Closure
Procedure: Delayed Primary Closure — A double antibiotic scheme with a cephalosporin and metronidazole is used as prophylaxis, and the fascia was closed with a continuous Polyglycolic Acid 0 suture. The wound is left open for at least 7 days, after which closure with Polypropylene 2-0 takes place if considered suitable by a board certified surgeon.
  Arms: Delayed Primary Closure

SUMMARY:
The objective of the study is to compare infection rates between primary, delayed primary and vacuum assisted closures in contaminated and dirty/infected laparotomy wounds.

DETAILED DESCRIPTION:
The objective of this study is to compare infection rates between primary, delayed primary and vacuum assisted closures in contaminated and dirty/infected laparotomy wounds.

Social, demographic, surgical, postsurgical and medical variables were registered. A descriptive analysis expressed as total and percentages, medians and interquartile ranges. Comparison between groups was made using the Kruskal-Wallis, U-Mann Whitney or Chi-squared as appropriate. A p value of less than 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Laparotomy wound classified as class III or IV according to CDC's Criteria for Defining a Surgical Site Infection.

Exclusion Criteria:

* Patient refusal to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Surgical Wound Infection with each Wound Closure Technique | Two months
  Presence of infection was determined by a certified board physician according to CDC's Criteria for Defining a Surgical Site Infection.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Lozano Balderas, MD, Principal Investigator — Escuela Nacional de Medicina, Tecnologico de Monterrey
Locations (1):
- Escuela Nacional de Medicina, Tecnologico de Monterrey, Monterrey, Nuevo León, Mexico